CLINICAL TRIAL: NCT05711134
Title: Audit and Feedback for Computed Tomography of the Cervical Spine in the Emergency Department
Brief Title: CT C-spine Audit and Feedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Karl Chamberlin, Assistant Professsor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY00000533
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Cervical Spine Injury; Emergencies; Trauma
Keywords: computed tomography; resource utilization; NEXUS; emergency medicine
MeSH Terms: conditions — Emergencies; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Serial In-Person Feedback (Experimental): Providers are given recurring individualized in-person feedback on their practice patterns.
  Interventions: Behavioral: Audit and Feedback on Individual Practice Patterns
- In-Person Feedback with Serial Electronic Feedback (Experimental): Providers are given one-time individualized in-person feedback on their practice patterns, followed by recurrent individualized electronic feedback.
  Interventions: Behavioral: Audit and Feedback on Individual Practice Patterns
- Control (No Intervention): Providers are not given any feedback on their practice patterns.

INTERVENTIONS:
Behavioral: Audit and Feedback on Individual Practice Patterns — Providers are given feedback on their practice patterns of ordering computed tomography of the cervical spine.
  Arms: In-Person Feedback with Serial Electronic Feedback; Serial In-Person Feedback

SUMMARY:
This is a prospective quality improvement study to assess the effect of using an audit-and-feedback process for emergency providers on utilization of computed tomography of the cervical spine. The objective of this study is to determine whether providing repeated individualized feedback on CT C-spine utilization to emergency providers alters their practice pattern and reduces overutilization. The investigators hypothesize that emergency providers who receive individualized feedback regarding their CT C-spine utilization on a regular basis will alter their practice pattern to reduce overutilization of this imaging study.

ELIGIBILITY:
Inclusion Criteria:

* Emergency medicine physician, nurse practitioner, or physician assistant
* Ordered at least 5 CT scans of the cervical spine on adult patients in the two-month pre-intervention period

Exclusion Criteria:

* Non-emergency providers
* Ordered few than 5 studies in the pre-intervention period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Percent NEXUS-Negative | 6 months
  Percentage of CT C-spine studies that an individual provider ordered on NEXUS-negative patients

SECONDARY OUTCOMES:
Number of Fractures | 6 months
  Number of cervical spine fractures identified on CT for patients who are NEXUS-negative
Clinically Significant Fractures | 6 months
  Number of cervical spine fractures identified on CT for patients who are NEXUS-negative that required procedural intervention, hospitalization, or prolonged immobilization
Number of CTs | 6 months
  Number of CT scans of the cervical spine ordered by each provider

CONTACTS AND LOCATIONS:
Overall Officials: Karl T Chamberlin, MD, Principal Investigator — University of Massachusetts Chan Medical School
Locations (1):
- University of Massachusetts Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No